CLINICAL TRIAL: NCT05802537
Title: Home-Based Exergame Program for Community-Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungdong University (Other)
Responsible Party: Principal Investigator, Kyeongjin Lee, Professor, Kyungdong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1041455-202302-HR-003-01
Record Dates: First submitted 2023-03-18; First posted 2023-04-06 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Exergaming; Frail Elderly

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group engaged in a home-based exergame program for 50 minutes per session, three times per week, for eight weeks. The program focused on enhancing lower extremity strength and balance.
  Interventions: Behavioral: Home-based exergame program
- Control group (Active Comparator): The control group participated in weekly online education sessions for 50 minutes over an eight-week period. The topics covered included fall prevention, musculoskeletal health, aging, and fracture risks. No physical exercise intervention was given.
  Interventions: Behavioral: Online education on fall prevention and musculoskeletal health management

INTERVENTIONS:
Behavioral: Home-based exergame program — The home-based exergame program was conducted using the Nintendo Switch and Ring Fit Adventure program at participants' homes. The program included a 10-minute warm-up, 30 minutes of main exercise, and a 10-minute cool-down, lasting a total of 50 minutes per session. Sessions were held three times per week for eight weeks. The exercises targeted lower extremity strength, balance, and flexibility and included yoga, leg exercises (e.g., squats, knee lifts), and other activities performed in a gamified virtual environment. Participants received guidance on using the console, and family members were involved to support proper execution of the exercises.
  Arms: Experimental group
Behavioral: Online education on fall prevention and musculoskeletal health management — The online education intervention consisted of weekly sessions conducted for 50 minutes over an eight-week period, focusing on fall prevention and musculoskeletal health management. Participants joined the sessions via a video-conference platform. The content covered education on aging, musculoskeletal disorders, fall prevention strategies, and understanding falls and fractures. These sessions aimed to enhance participants' awareness and knowledge, thereby helping them adopt preventive behaviors.
  Arms: Control group

SUMMARY:
The purpose of this study was to investigate the effect of a home-based exergame program on physical function, fall efficacy, depression, and quality of life in older adults. For the purpose of the study, the investigators established the following hypotheses. Older adults who participate in a home-based exergame program will experience significant improvements in physical function, fall efficacy, depression, and quality of life compared to those who do not participate in the program.

ELIGIBILITY:
Inclusion Criteria:

* 75 years or older
* the ability to walk independently with or without a walking aid
* a mini-mental state examination score ≥ 24.

Exclusion Criteria:

* musculoskeletal disorders such as fractures or dislocations
* neurological impairment
* mental disorders
* uncontrolled endocrine, cardiovascular, or urinary system diseases

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
One-leg standing test | Change from baseline after intervention at 8 weeks
  The one-leg standing test was used to evaluate static postural balance. The one-leg standing test is a simple, reliable, and valid test for assessing balance and fall risk in older adults.
Berg balance scale | Change from baseline after intervention at 8 weeks
  To evaluate dynamic postural balance, the Berg balance scale was used. It has a perfect score of 56 and consists of 14 items, with a perfect score of 4 for each item.
Functional reaching test | Change from baseline after intervention at 8 weeks
  Functional reaching test was used to evaluate movement limits.
Timed up-and-go test | Change from baseline after intervention at 8 weeks
  Timed up-and-go test was used to assess functional movement and mobility.
Five-times sit-to-stand test | Change from baseline after intervention at 8 weeks
  Five-times sit-to-stand test was used to evaluate lower-extremity muscle strength.

SECONDARY OUTCOMES:
Falls Efficacy | Change from baseline after intervention at 8 weeks
  Falls efficacy was evaluated using the Modified Falls Efficacy Scale (MFES), which was specifically developed for older adults. The MFES consists of 14 questions, each scored from 0 (not confident) to 10 (very confident). The total score ranges from 0 to 140, with higher scores indicating greater confidence in performing activities without falling, which is considered a better outcome.
Depression | Change from baseline after intervention at 8 weeks
  Depression was measured using the Geriatric Depression Scale-15 (GDS-15), a validated screening tool for older adults. The GDS-15 consists of 15 yes/no questions, with scores ranging from 0 to 15. Higher scores represent more severe depressive symptoms, which is considered a worse outcome.
Health-Related Quality of Life | Change from baseline after intervention at 8 weeks
  Health-related quality of life was measured using the 36-Item Short Form Health Survey (SF-36), which assesses multiple domains of health status, including physical functioning, pain, role limitations, emotional problems, mental health, social functioning, vitality, and general health. The SF-36 contains 36 items, each rated on a scale from 1 to 5, with the total score converted to a range from 0 to 100. Higher scores indicate better health outcomes, reflecting a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kyungdong University, Wŏnju, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee K. Home-Based Exergame Program to Improve Physical Function, Fall Efficacy, Depression and Quality of Life in Community-Dwelling Older Adults: A Randomized Controlled Trial. Healthcare (Basel). 2023 Apr 12;11(8):1109. doi: 10.3390/healthcare11081109. PMID 37107943